CLINICAL TRIAL: NCT00005616
Title: A Phase I Single Dose-Escalation Study of BIBH-1 in Patients With Colorectal Cancer Scheduled for Surgical Resection
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-035A; CDR0000067753 (Registry Identifier: PDQ (Physician Data Query)); BOEH-1152.5; LUDWIG-LUD98-006; NCI-G00-1756
Record Dates: First submitted 2000-05-02; First posted 2004-06-18 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Neoadjuvant Therapy

INTERVENTIONS:
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Procedure: radionuclide imaging
Radiation: iodine I 131 monoclonal antibody F19

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of monoclonal antibody therapy in treating patients who have colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine any toxicity associated with increasing single doses of monoclonal antibody F19 (BIBH-1) administered by intravenous infusion in patients with colorectal cancer scheduled for surgical resection. II. Compare the pharmacokinetics, biodistribution, and imaging characteristics of increasing intravenous doses of iodine I 131 BIBH-1 in this patient population. III. Compare the BIBH-1 related human antihuman antibody (HAHA) serum concentration with immunologic related clinical effects in these patients. IV. Compare the uptake of iodine I 131 BIBH-1 in tumor to the uptake of normal tissue when administered to these patients.

OUTLINE: This is a dose escalation study. Patients receive monoclonal antibody F19 (BIBH-1) combined with iodine I 131 IV over 60 minutes. Patients undergo surgical resection approximately 7 days after BIBH-1 infusion. Cohorts of 3-6 patients receive escalating doses of BIBH-1 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities. Patients are followed once during days 5-14 and then at day 30 after surgery.

PROJECTED ACCRUAL: A total of 12 patients will be accrued for this study within 4 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed primary colorectal cancer Candidate for a clinically indicated laparotomy for primary tumor resection, resection of hepatic metastases, or placement of an intrahepatic arterial catheter No active CNS metastases defined by new or enlarging lesions on CT scan or within 3 months of treatment (i.e., surgery or radiotherapy) for brain metastases No prior participation in this study

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: At least 3 months Hematopoietic: Granulocyte count at least 2,500/mm3 Lymphocyte count greater than 700/mm3 Platelet count at least 100,000/mm3 Hepatic: ALT/AST no greater than 3 times upper limit of normal Bilirubin less than 2 mg/dL Renal: Creatinine no greater than 2.0 mg/dL Other: No pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No incomplete healing at an incision site as evidenced by incomplete granulation, infection, or localized edema No active infections requiring antibiotics No bleeding disorders No other serious illness that may potentially interfere with obtaining accurate study results No autoimmune disease No hypertrophic skin conditions

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy No prior murine, chimeric, or humanized antibody and/or antibody fragment Chemotherapy: At least 4 weeks since prior chemotherapy Endocrine therapy: No concurrent systemic corticosteroids except for acute management of allergic type events Radiotherapy: See Disease Characteristics Surgery: See Disease Characteristics Recovered from prior surgery Other: At least 4 weeks since other prior investigational agents No concurrent immunosuppressive agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 1999-09; Primary Completion 2000-08 (Actual); Study Completion 2000-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sydney Welt, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States